CLINICAL TRIAL: NCT01939860
Title: A Feasibility Study of the Impact on Blood Pressure Control of Supplementing Community Pharmacist Services With Structured Information on Blood Pressure and Its Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Responsible Party: Principal Investigator, Ejaz Cheema, PhD student, University of Warwick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Warwick.123
Record Dates: First submitted 2013-09-03; First posted 2013-09-11 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual pharmacy care (No Intervention): Participants will not receive any structured written education on hypertension and its treatment
- usual pharmacy care plus structured information (Experimental): Participants will be provided with validated verbal and written information on hypertension and its treatment, including information about class (es) of anti-hypertensive medication(s) used by each patient, and their common side-effects. The written material will be based on validated patient information leaflets from the British Heart Foundation and the Blood Pressure Association.
  Interventions: Other: Written and verbal patient education on hypertension and its treatment

INTERVENTIONS:
Other: Written and verbal patient education on hypertension and its treatment
  Arms: usual pharmacy care plus structured information

SUMMARY:
Hypertension is a major health problem, however its control is unsatisfactory. One of the reasons for such a high prevalence of this disease includes poor patient compliance to treatment. Approximately 30 % of newly diagnosed hypertensive patients stop taking their blood pressure medication by six months and 50% by 12 months.

The UK government is keen to encourage community pharmacists to play an active role in participation of services that can improve patient adherence to their medications. The New Medicines Service (NMS) and targeted Medicines Use Reviews (MUR) are established services which fund community pharmacists to review and explain medicine use to patients, with hypertension a common condition for which advice is given within these schemes. Within these schemes, advice is verbal and unstructured, with no specific written information provided on drugs or the disease being treated.

This study aims to determine whether structured information provided to participants verbally and in writing by community pharmacists about blood pressure and current medicine(s) within NMS and targeted MURs will be retained and will be associated with improved hypertension control. Participants will be recruited from people eligible for NMS and MURs and attending community pharmacies.

ELIGIBILITY:
Inclusion Criteria:

1)18 or over 2) male or female 3) Have been started on any blood pressure medication

Exclusion Criteria:

1)Patients with English language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in systolic or diastolic blood pressure | 1 year (trial would be stopped at 26 weeks if it is not possible to recruit any further participants
  Systolic and diastolic blood pressure will be measured and recorded in mm Hg using OMRON blood pressure monitors

SECONDARY OUTCOMES:
change in the knowledge of hypertension | one year(trial would be stopped at 26 weeks if it is not possible to recruit any further participants)

CONTACTS AND LOCATIONS:
Locations (1):
- J P Goes chemist, Coventry, United Kingdom